CLINICAL TRIAL: NCT05792345
Title: Comparison of Post-operative Analgesia in Pediatric Superficial TTMPB
Acronym: PEPOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Professor, MD, Priva Docent, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEPOST 2022-01964
Record Dates: First submitted 2023-02-23; First posted 2023-03-31 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Regional Anesthesia
Keywords: regional anesthesia; pediatric; cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Infiltration will be performed by surgeon at the site of sternotomy
  Interventions: Procedure: Control
- With TTMPB (Active Comparator): Regional anesthesia is performed with direct view of the nerves and vascular position
  Interventions: Procedure: Transversus Thoracic Muscle Plane Block

INTERVENTIONS:
Procedure: Transversus Thoracic Muscle Plane Block — The transversus thoracic muscle plane block It is most commonly performed following cardiothoracic surgeries (or any surgeries requiring sternotomy) to provide analgesia to the anterior chest wall. he TTMPB, and thoracic fascial plane blocks, are increasingly being employed as part of enhanced recovery after surgery (ERAS) protocols for cardiothoracic procedures. They have been shown to significantly reduce both the time to extubation and the incidence of acute and chronic perioperative pain
  Arms: With TTMPB
Procedure: Control — Infiltration by surgeon
  Arms: Control

SUMMARY:
When a patient is to undergo heart surgery with a sternotomy, a transthoracic block is performed. The thoracic block is an analgesic technique which consists of injecting anesthetic product into the nerves, in order to avoid significant pain. The common technique is to make injections in the sternum by the surgeon. A new, increasingly widespread method is performed by the anesthetist who performs the block under ultrasound.

This research project aims to determine if performing this transthoracic block under ultrasound is more effective than injections performed by the surgeon without ultrasound.

DETAILED DESCRIPTION:
Cardiac surgery, and more specifically associated sternotomy, leads to severe pain in the postoperative period. Adequate analgesia is therefore challenging, but of paramount importance to reduce associated side effects such as pulmonary hypertensive crisis, tachyarrhythmia, systemic hypertension, hypoxia, and increased morbidity and length of stay. Actual opioid crisis and risks associated with intravenous analgesics raises the question of having an alternative and better approach to relieve severe pain. Currently in the postoperative suites opiates are also used for sedative purposes. This strategy of sedation has to change. Recent advances in regional anaesthesia could be the answer.

Thoracic epidural or paravertebral blocks provide effective analgesia for open cardiac surgery in paediatric patients. However, the major risk of epidural hematomas caused by heparinization, hemodynamic instability, technical difficulties and pneumothorax has limited the application of these two techniques in open cardiac surgery, and promoted the development of new approaches with safe, reliable, and cost-effective techniques, such as ultrasound-guided peripheral nerve blocks. This might be the most effective method for pain management in paediatric patients undergoing cardiac surgery according to recent studies. Superficial Thoracic Transversus Muscle Plane Block has been recently described and evaluated for pain management in adult cardiac surgery. It works through the blockade of multiple anterior branches of the intercostal nerves (Th2-6) in the internal mammary region. It has also been described in children in a few papers: Zhang and al. in a randomized controlled trial in 100 children, Abdelbaser and al. conducted a randomized double blind study including 80 children. In these studies, the injection of local anaesthetics was made between the intercostal and transversus thoracis muscles. But in very small children, the risk of pleura or internal mammary artery puncture associated with this injection is relatively important. Superficial TTMPB (located between the intercostal and pectoralis major muscles) seems to have the same analgesic potency without the aforementioned risks.That is to say that TTMPB is better than nothing but, to our knowledge, there is no study comparing infiltration by surgeon and TTMPB.

The risks of the procedure are the same with all regional anaesthesia, which are vascular or nerves punction, hematoma and failure of anaesthesia.

This study is set up to test the hypothesis that analgesia performed by TTMPB may have a better antalgic effect than blocks made by surgeons, in patients who undergo cardiac sternotomy. At first, the standard in CHUV was injections made by surgeon. Nowadays the decision of technic used is made with a discussion between anesthesist and surgeon during operative time. The investigators want to bring an evidence based decision with this study.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing sternotomy for a cardiac surgery in CHUV, which is an academic hospital in Switzerland.

Participants fulfilling all of the following inclusion criteria are eligible for the study :

* Informed Consent as documented by signature.
* Age from 0 to 16 years old.
* Undergoing cardiac surgery with sternotomy in CHUV, Lausanne.

Exclusion Criteria:

* • Patients older than 16 years.

  * Pregnancy.
  * Sternotomy for operation other than cardiac surgery.
  * Contraindication to local anesthesic, e.g. known hypersensitivity or allergy to Bupivacaine.
  * Infection at the site of injection.
  * Not having consented for this procedure/ refusal of participation. Reoperation during the same hospitalisation.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Opioids dose | Day 0, Hour 24 post-operative.
  Opioids dose administered for analgesia in mg and divided by patient weight in kg

SECONDARY OUTCOMES:
Opioids dose | Day 0 at Hour 4, 12 and Day 1 post-operative
  Opioids dose administered for analgesia in mg and divided by patient weight in kg
Time to extubation | From the time of arrival in the Intensive Care Unit until the time of extubation assessed up to 3 months
  Time to extubation in minutes
Dose of catecholamine (noradrenaline) used | At Day 0 Hour 4, 12, 24 and Day 1 post-operative
  Total dose per kg infused
Length of stay in ICU before discharge | From the time of arrival in the Intensive Care Unit until discharge assessed up to 3 months
  Length of stay in ICU before discharge in days
Adverse Event | Day 1 post operatively
  Analysis of adverse events and adverse events of special interest (complications) such as hematomas, arterial puncture, fail of the block, pneumothorax.
FLACC pain scale (Face, Legs, Activity, Cry, Consolability) | at Day 0 at Hours 4, 12 and 24 post-operative;
  Postoperative pain evaluated by the Flacc pain scale, From 0 to 10 were 10 is the worst pain experimented by the patient and 0 is the normal state.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Mauron, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bettex DA, Schmidlin D, Chassot PG, Schmid ER. Intrathecal sufentanil-morphine shortens the duration of intubation and improves analgesia in fast-track cardiac surgery. Can J Anaesth. 2002 Aug-Sep;49(7):711-7. doi: 10.1007/BF03017451. English, French. PMID 12193491
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179
- [Background] Ueshima H, Kitamura A. Blocking of Multiple Anterior Branches of Intercostal Nerves (Th2-6) Using a Transversus Thoracic Muscle Plane Block. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):388. doi: 10.1097/AAP.0000000000000245. No abstract available. PMID 26079353
- [Background] Zhang Y, Chen S, Gong H, Zhan B. Efficacy of Bilateral Transversus Thoracis Muscle Plane Block in Pediatric Patients Undergoing Open Cardiac Surgery. J Cardiothorac Vasc Anesth. 2020 Sep;34(9):2430-2434. doi: 10.1053/j.jvca.2020.02.005. Epub 2020 Feb 11. PMID 32151511
- [Background] Abdelbaser II, Mageed NA. Analgesic efficacy of ultrasound guided bilateral transversus thoracis muscle plane block in pediatric cardiac surgery: a randomized, double-blind, controlled study. J Clin Anesth. 2020 Dec;67:110002. doi: 10.1016/j.jclinane.2020.110002. Epub 2020 Jul 24. PMID 32717448
- [Background] Ohgoshi Y, Ino K, Matsukawa M. Ultrasound-guided parasternal intercostal nerve block. J Anesth. 2016 Oct;30(5):916. doi: 10.1007/s00540-016-2202-5. Epub 2016 Jun 20. No abstract available. PMID 27325411